CLINICAL TRIAL: NCT00146666
Title: Evaluation of FM220 in Patients With Peripheral Arterial Disease (PAD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: FlowMedic (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05US01
Record Dates: First submitted 2005-09-03; First posted 2005-09-07 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-08

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peak walking time; Absolute claudication distance; Claudication onset time; Initial claudication distance; Intermittent compression
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Intermittent Pneumatic Compression Devices

INTERVENTIONS:
Device: Intermittent compression

SUMMARY:
The purpose of this study is to determine whether 12 weeks of daily home use of the FM220 in the most affected leg of patients with PAD and claudication, will improve peak walking time (PWT) at three months as compared with a non-treated control group.

ELIGIBILITY:
Inclusion Criteria(main):

1. Patients aged 40 or more.
2. Peripheral arterial disease as determined by resting ABI<0.90.
3. Reduction in post exercise Ankle Brachial Index (ABI) of > 20% in the symptomatic limb.
4. Stable claudication for the past three months
5. Baseline PWT between 1 and 10 minutes
6. If the patient is under claudication drug therapy (eg. cilostazol and pentoxifvlline) the use and dose of these drugs has been stable for the last 60 days.
7. If the patient is receiving of statin and antiplatelet therapy, the use and dose of these drugs has been stable for the last 60 days.

Exclusion Criteria:

1. Any active pathological heart, muscular, neurological, orthopedic, cognitive or pulmonary disease which might interfere with patient compliance or ability to walk on a treadmill in the opinion of the investigator.
2. Non compressible arteries as defined by ABI>1.1
3. Clinical evidence of acute or subacute superficial or deep venous thrombosis confirmed by continuous-wave Doppler in the affected extremity.
4. Deep venous insufficiency on clinical grounds or by lab measurements.
5. Prior below-knee surgical revascularization procedure within the last 6 months.
6. Significant likelihood of lower extremity arterial revascularization procedure within the next 6 months.
7. Ulcer, cellulitis, skin conditions, or superficial thrombophlebitis in regions covered by the compression device preventing use of the device.
8. Acute pulmonary embolism.
9. Osteomyelitis of the lower extremity.
10. Gangrene of the lower extremity.
11. Acute limb ischemia.
12. Clinical scenarios in which increased venous or lymphatic return is undesirable.
13. Painful calf conditions which would exclude use of the pump.
14. Peripheral neuropathy that, in the opinion of the investigator, would prevent patient from accurately assessing claudication symptoms or identifying Cutaneous comfort of the device Vein ligation.
15. Pulmonary edema.
16. Significant aorto-iliac disease as demonstrated by physical examination or objective testing. Absence of aorto-iliac disease must be documented by segmental testing performed within 90 days of study enrollment.
17. Critical leg ischemia with evidence of rest pain, ischemic ulceration, gangrene.
18. Participation in any clinical trial within the past 30 days.
19. Morbid obesity, defined by BMI>40, weight greater than 300 lbs or leg circumference greater than 19.7 inches.
20. Pregnancy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-09; Study Completion 2006-09 (Estimated)

PRIMARY OUTCOMES:
Increase in Peak Walking Time as determined on graded treadmill test at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koren, MD, Principal Investigator — Jacksonville Center For Clinical Research; Jeffrey M Martinez, MD, Principal Investigator — Peripheral Vascular Associates
Locations (2):
- United States (2):
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Peripheral Vascular Associates, San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.flowmedic.com/